CLINICAL TRIAL: NCT02533479
Title: Erythrocytes and Skeletal-muscle Unsaturated and Omega-6 Fatty Acids Are Positively Correlated After Caloric Restriction and Exercise
Brief Title: Erythrocytes and Skeletal-muscle Fatty Acids Are Positively Correlated After Caloric Restriction and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Alt Rendiment (Other)
Responsible Party: Principal Investigator, FRANCISCO DROBNIC, MD, PhD, PhD in Medicine, Centre d'Alt Rendiment
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAR-1
Record Dates: First submitted 2015-07-07; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Caloric restriction (Experimental): three alternate days weekly along 4 weeks.
  Interventions: Other: Caloric restriction

INTERVENTIONS:
Other: Caloric restriction — three alternate days weekly along 4 weeks.

SUMMARY:
The aim is compare and correlate skeletal muscle and erythrocytes fatty acids (FAs) profiles in adult healthy human after caloric restriction and acute exercise in order to validate erythrocyte FAs profile as marker of changes in muscle fatty acid composition.

DETAILED DESCRIPTION:
The study was performed with 11 healthy sportsmen participating in a caloric restriction trial for 1 month. The participants follow a caloric restriction, 30-40% respect to the usual diet of each participant, three alternate days weekly along 4 weeks. After the caloric restriction period the participants realized an exercise stress test. For each participant one blood sample and muscular biopsy were obtained after acute exercise and caloric restriction intervention. All the participants were informed of the purpose and demands of the study before giving their written consent to participate. The study protocol was in accordance with the Declaration of Helsinki for research on human participants and was approved by the local Ethics Committee of the Consell Català de l'Esport.

ELIGIBILITY:
Inclusion Criteria:

* age (18-50 years old),
* sex (male),
* equilibrate diet and physical activity of 3 days weekly.

Exclusion Criteria:

* sex (female),
* smokers.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in skeletal muscle FAs profiles in adult healthy human after caloric restriction and acute exercise | 8 weeks
  Muscular biopsy was obtained from vastus lateralis of the quadricipitalis muscle. The dermis was cut for to display muscular aponeurosis (<2.5 cm) after clean and sterilize the biopsy zone. Next the aponeurosis was cut and a puncture with Vacora® device (Bard Biopsy Systems, Tempe, AZ, USA) was realized. The injury was cleaned and sutured, and the muscular sample was stored at -80ºC until FA analyses..FA composition of skeletal muscle were determined by gas chromatography.
Changes in erythrocytes FAs profiles in adult healthy human after caloric restriction and acute exercise | 8 weeks
  Venous blood samples were obtained from the antecubital vein of participants with vacutainers containing EDTA (ethylenediaminetetraacetic acid) as anticoagulant (6 mL) to purify erythrocytes following an adaptation of the method described elsewhere (Boyum, 1964; Sureda et al., 2006). Erythrocyte fraction was obtained after centrifugation (900 x g, 30 min, 4ºC). Then, erythrocytes were cleaned with phosphate buffered saline (PBS), centrifuged (900 x g, 20 min, 4ºC) and lysed with water at initial blood volume. Cell lysates were stored at -80ºC until FA analyses. FA composition of erythrocytes were determined by gas chromatography.

SECONDARY OUTCOMES:
Densitometry | 8 weeks
  Densitometry was performed by Lunar IDXA (General Electric, USA)
Exercise stress test energy efficiency | 8 weeks
  Standardized maximal treadmill exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Franchek Drobnic, Ph D, Study Chair — Centre d'Alt Rendiment, Sant Cugat
Locations (1):
- Centre D'Alt Rendinemt, Sant Cugat, Barcelona, Spain

REFERENCES:
- [Background] Capo X, Martorell M, Sureda A, Tur JA, Pons A. Effects of docosahexaenoic supplementation and in vitro vitamin C on the oxidative and inflammatory neutrophil response to activation. Oxid Med Cell Longev. 2015;2015:187849. doi: 10.1155/2015/187849. Epub 2015 Apr 19. PMID 25960826
- [Derived] Pons V, Riera J, Capo X, Martorell M, Sureda A, Tur JA, Drobnic F, Pons A. Calorie restriction regime enhances physical performance of trained athletes. J Int Soc Sports Nutr. 2018 Mar 9;15:12. doi: 10.1186/s12970-018-0214-2. eCollection 2018. PMID 29556158